CLINICAL TRIAL: NCT03515291
Title: A Phase IIB, Randomised, Double-Blinded, Placebo-Controlled Study of the Efficacy and Safety of Intramyocardial Injection of Allogeneic Human iMP Cells in Patients Undergoing CABG Surgery.
Brief Title: A Trial of Cardiac Injections of iMP Cells During CABG Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cell Therapy Ltd. (Industry)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLX003-IMP-2-170121
Record Dates: First submitted 2018-04-20; First posted 2018-05-03 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Myocardial Fibrosis
Keywords: Heart; CABG; Injection; Scar; Fibrosis; Cell; Progenitor; Immunomodulatory; MRI; Randomized
MeSH Terms: conditions — Cicatrix; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- iMP cell injection (Experimental): iMP cells injected in to the epicardial surface of the heart during coronary artery bypass graft surgery.
  Interventions: Biological: iMP cells
- Control injection (Placebo Comparator): Control (cell suspension solution) injected in to the epicardial surface of the heart during coronary artery bypass graft surgery.
  Interventions: Other: Control injection

INTERVENTIONS:
Biological: iMP cells — Immunomodulatory progenitor cells
  Other Names: "Heartcel"
  Arms: iMP cell injection
Other: Control injection — Cell suspension solution
  Arms: Control injection

SUMMARY:
Injury to the heart, which may occur following a heart attack or owing to the mechanical effect of high blood pressure, leads to scarring (fibrosis) of the heart muscle. Fibrosis of the muscle can cause impaired pumping of the heart, which can lead to heart failure, and the abnormal conduction of electrical signals through the heart. This may in turn lead to abnormal, potentially fatal, heart rhythms. Currently, scarring of the heart muscle cannot be reversed and is generally progressive.

A previous clinical study found that participants who received injections of immunomodulatory progenitor cells (iMP cells, "Heartcel") showed a reversal of heart muscle scarring when the cells were injected into heart muscle during coronary artery bypass graft (CABG) surgery. However, the previous trial was a small scale study and did not have a control group. The aim of this study is to perform a larger scale investigation with 50 participants compared to the previous trial of 11, and split the 50 participants into two groups - a test group and a control group, so that a direct comparison may be made between the two groups.

DETAILED DESCRIPTION:
Myocardial fibrosis is a currently untreatable medical condition. A previous trial reported that when iMP cells, a cell type of mesodermal lineage which is separate from, but shares characteristics with, mesenchymal stem cells (MSCs), were injected into the myocardium during CABG surgery, there was a reduction in the degree of scarring relative to baseline observed on 4 month and 12 month Single-Photon Emission Computed Tomography (SPECT) images.

The previous trial was open label with 11 participants and no control group, only historic comparisons. The proposed trial will be larger and will include a control group. The trial endpoints have been updated to take account of the findings of the first trial and late gadolinium enhanced (LGE) Magnetic Resonance Imaging (MRI) scans (LGE-CMR), which have higher resolution than SPECT scans, will be used to assess the appearance of fibrosis.

iMP cells were developed by the sponsor as an allogeneic mesodermally derived cellular therapy for cardiac conditions. While iMPs are plastic adherent like MSCs, iMPs do not meet the International Society for Cellular Therapy's definition of MSCs, though like MSCs, markers indicate that iMPs are immune privileged and can therefore be employed allogeneically without inducing a significant immune response.

The trial is open to participants, male and female, who require CABG surgery and have 15% or greater left ventricular scarring. Unless part of normal clinical care, participants will be required to undergo a screening LGE-MRI to assess the degree of left ventricular scarring. The MRI however, may reveal that the individual is not eligible to participate in the study. If the individual is eligible, then the LGE-MRI will be used as the baseline recording and to plan the injection sites.

Each participant will be involved in the study for approximately 4.5 months. There will be two outpatient pre-operative hospital visits which will occur up to 6 weeks prior to surgery, though if a potential participant is an inpatient, the pre-operative eligibility/baseline tests can be performed over a shorter period of time as an inpatient. The CABG surgery will not differ from normal, except for the injections into the heart muscle, and participants will not miss out on any standard care. There will then be follow up visits at 1 week, 1 month and 15±2 weeks post surgery. The 1 week visit may occur as an inpatient depending on post-operative improvement. The follow up visits will not involve overnight stays. Follow up visits will mainly entail an ECG, an echocardiogram, a blood test, a urine test, health questionnaires and a discussion about the participant's health and any adverse events. Specific details are available from the chief investigator, see below. The 15±2 week visit will also involve a follow up LGE-MRI for primary endpoint assessment. After this visit, participation in the study will end and participants will receive only the normal post CABG care.

As this is a quadruple blind randomised controlled trial, neither participants nor care staff will know to which group a participant is allocated. Of the 50 participants, 30 will receive injections of cells and 20 will receive control injections.

ELIGIBILITY:
Inclusion Criteria:

Greater than or equal to 15% LV scar volume measured by LGE-CMR.

LVEF ≤50%.

Ischaemic heart disease where CABG is the recommended revascularisation strategy.

Age range: 18 years of age and over with no history of congenital cardiac anomalies (men and women).

Able to provide written informed consent (including willingness to have two CMRs).

New York Heart Association (NYHA) class >=2 and/or Canadian Cardiovascular Society (CCS) class angina >=2.

For women of child bearing potential (WOCBP): Negative (non-pregnant) beta-human chorionic gonadotropin (beta-hCG) blood test.

Exclusion Criteria:

Previous cardiac surgery

Requirement for additional cardiac surgery including concomitant valve replacement surgery.

Estimated GFR of <30mL/min

Contraindication to performance of CMR

Clinical history of malignancy within 5 years

Comorbidities likely to influence the safety of performing the protocol

Liver disease including ALT 3 times or more the upper limit of normal

Low platelet count (<100,000) platelets per microliter of blood

Evidence of coagulopathy - International Normalised Ratio (INR) >2. Note: Elevated INR due solely to warfarin (or similar medication) is NOT an exclusion criterion.

Increased mortality risk over a 12-month period due to comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants must not be pregnant (negative beta hCG test).
Enrollment: 50 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
LGE-CMR | Baseline and 15±2 weeks post surgery
  Change in left ventricular LGE-CMR imaging (e.g. scar/fibrosis volume reduction), iMP group compared to control group.

SECONDARY OUTCOMES:
LGE-CMR | Baseline and 15±2 weeks post surgery
  Difference in Left Ventricular Ejection Fraction (LVEF), Left Ventricular End-Diastolic Volume Index (LVEDVi), Left Ventricular End-Systolic Volume Index (LVESVi), LV late gadolinium enhancement pattern, myocardial perfusion and myocardial strain.
Major Adverse Cardiac Events (MACE) | Recorded 1 month and 15±2 weeks post surgery
  Comparison of MACE rates between the two groups - Cardiovascular death, non fatal MI, non fatal stroke and unplanned cardiovascular hospitalisation.
Major arrhythmic events | Recorded 1 month and 15±2 weeks post surgery
  Comparison of rates between the two groups.
All cause mortality | Recorded 1 month and 15±2 weeks post surgery
  Comparison of rates between the two groups.
New York Heart Association (NYHA) Class | Baseline and 15±2 weeks post surgery
  Assessment of difference in NYHA class between groups.
Quality of life questionnaires | Baseline and 15±2 weeks post surgery
  Kansas City Cardiomyopathy Questionnaire (KCCQ), the Minnesota Living with Heart Failure (MLHF) questionnaire and the EQ5D questionnaire - compared between the two groups.
Length of stay in intensive care/high dependency unit and time to discharge | Operation date until discharge from hospital date, assessed up to 30 days post surgery.
  Comparison of length of stay in intensive care/high dependency unit and time to discharge - compared between the two groups.
Blood biomarkers (routine and exploratory) | Baseline, 4 times during the post operative recovery period (12h, 24h, 48h and 72h) and at 1 week, 30 days and 15±2 weeks post surgery.
  Blood biomarkers related to cardiac function. Routine - Urea and electrolytes, liver function tests and full blood count. Exploratory - Uric acid, lipid profile, high sensitivity C reactive protein, high sensitivity troponin, N terminal pro brain natriuretic peptide. Levels compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Scott, MB BChir PhD, Study Director — Cell Therapy Ltd.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anastasiadis K, Antonitsis P, Westaby S, Reginald A, Sultan S, Doumas A, Efthimiadis G, Evans MJ. Implantation of a Novel Allogeneic Mesenchymal Precursor Cell Type in Patients with Ischemic Cardiomyopathy Undergoing Coronary Artery Bypass Grafting: an Open Label Phase IIa Trial. J Cardiovasc Transl Res. 2016 Jun;9(3):202-213. doi: 10.1007/s12265-016-9686-0. Epub 2016 Apr 1. PMID 27037806